CLINICAL TRIAL: NCT03717168
Title: Role of Recombinant Human Growth Hormone rHGH in Weaning of Prolonged Ventilation After Major Abdominal Cancer Surgeries.
Brief Title: Effects of Growth Hormone on Difficult Ventilator Weaning Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Principal investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ehab- Mahmoud growth hormone
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Mechanical Ventilation Complication
Keywords: recombinant growth hormone; Difficult ventilator weaning; postoperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Growth Hormone; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant human growth hormone (Active Comparator): Patients who received growth hormone immediately after tracheostomy.
  Interventions: Drug: Recombinant human growth hormone
- Control (Active Comparator): Patients who did not receive growth hormone and followed the conventional weaning trials
  Interventions: Other: Control

INTERVENTIONS:
Drug: Recombinant human growth hormone — All the patients received subcutaneous rHGH (0.3 IU/kg/ twice daily) for 10 days in addition to intensive care standard management.
  Other Names: drug group
  Arms: Recombinant human growth hormone
Other: Control — All patients will not receive growth hormone.
  Other Names: control group
  Arms: Control

SUMMARY:
Major abdominal surgeries may be followed by postoperative pulmonary complications (PPCs). These complications are common and can cause significant morbidity and mortality.

Major operations are followed by acute respiratory insufficiency (RI) in 3%-27.4%, which causes prolonged hospital stay, high patient costs, high mortality rate and lower survival rates. The most crucial pulmonary postoperative complication is the prolonged mechanical ventilation and difficult weaning.The rHGH is a synthetic metabolic hormone which improves synthesis of protein, corrects hypoalbumenia, reverses negative nitrogen balance, improves patient nutrition, improves wound healing and promotes recovery of respiratory muscle function. When used for weaning from mechanical ventilation, rHGH reducess the duration of mechanical ventilation time, ICU admission period, incidence of VAP & ICU mortality.

DETAILED DESCRIPTION:
Major abdominal surgeries may be followed by postoperative pulmonary complications (PPCs). These complications are common and can cause significant morbidity and mortality.

Major operations are followed by acute respiratory insufficiency (RI) in 3%-27.4%, which causes prolonged hospital stay, high patient costs, high mortality rate and lower survival rates. The most crucial pulmonary postoperative complication is the prolonged mechanical ventilation and difficult weaning.The rHGH is a synthetic metabolic hormone which improves synthesis of protein, corrects hypoalbumenia, reverses negative nitrogen balance, improves patient nutrition, improves wound healing and promotes recovery of respiratory muscle function. When used for weaning from mechanical ventilation, rHGH reducess the duration of mechanical ventilation time, ICU admission period, incidence of VAP & ICU mortality. Felbinger et al reported a case of prolonged ventilation with failure of weaning after 42 days; the patient received subcutaneous rHGH (0.3 IU/kg/day) for 20 days in addition to intensive care standard management. They reported improvement of protein metabolism in addition to improvement of respiratory muscle strength, the patient was weaned successfully on the 75th postoperative day.this study assumes a hypothesis that rHGH would help weaning from mechanically ventilated tracheostomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major abdominal cancer surgeries.
* Patients requiring prolonged postoperative ventilation.
* Patients with multiple failed trials of mechanical ventilation weaning.
* ASA I and II patients.

Exclusion Criteria:

* History of chronic cardiac,renal or respiratory illness.
* Septic or septic shock patients on inotropic supports.
* Fully alert and Conscious patients.
* ASA 3 and 4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
The effect of rHGH on the mechanical ventilation time in patients underwent abdominal cancer surgery and needed postoperative mechanical ventilation for a long period | up to 6 weeks.
  The total mechanical ventilation days.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
after finishing the study and submitting to a highly impact journal will share the data and results.

REFERENCES:
- See also: the use of growth hormone for postoperative respiratory failure — https://www.ncbi.nlm.nih.gov/pubmed/8678203